CLINICAL TRIAL: NCT05228028
Title: Suprainguinal Fascia Iliaca Compartment Block Versus Anterior Quadratus Lumborum Block for Analgesia After Total Hip Arthroplasty: a Randomized Controlled Trial
Brief Title: Fascia Iliaca Compartment Block Versus Quadratus Lumborum Block in Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Seokha Yoo, Clinical Assistant Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2112-062-1282
Record Dates: First submitted 2022-01-18; First posted 2022-02-08 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Nerve Block; Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fascia iliaca compartement block [FICB] group (Experimental)
  Interventions: Procedure: fascia iliaca compartement block
- quadratus lumborum block [QLB] group (Experimental)
  Interventions: Procedure: quadratus lumborum block

INTERVENTIONS:
Procedure: fascia iliaca compartement block — Ultrasound-guided suprainguinal FICB (30 ml of 0.375% ropivacaine with 75 µg of epinephrine) is done on the ipsilateral surgical side at the end of surgery.
  Other Names: FICB
  Arms: fascia iliaca compartement block [FICB] group
Procedure: quadratus lumborum block — Ultrasound-guided anterior QLB (30 ml of 0.375% ropivacaine with 75 µg of epinephrine) is done on the ipsilateral surgical side at the end of surgery.
  Other Names: QLB
  Arms: quadratus lumborum block [QLB] group

SUMMARY:
Patients undergoing total hip arthroplasty are randomly assigned to two groups (fascia iliaca compartement block [FICB] group or quadratus lumborum block [QLB] group). In the FICB group, ultrasound-guided suprainguinal FICB (30 ml of 0.375% ropivacaine with 75 µg of epinephrine) is performed on the ipsilateral surgical side at the end of surgery. In the QLB group, ultrasound-guided anterior QLB (30 ml of 0.375% ropivacaine with 75 µg of epinephrine) is done on the ipsilateral surgical side at the end of surgery. A standardized multimodal analgesic regimen is used for postoperative pain control. The total use of opioids including patient-controlled analgesia and rescue analgesics is compared in both groups for 24 hours after surgery. The amount of opioids used is compared by conversion to oral morphine equivalent dose. Pain score at rest and movement during postoperative 24 hours, time to first request for analgesics, the incidence of side effects, patient satisfaction for pain control at postoperative 24 hours, quality of recovery at postoperative 24 hours, time to discharge readiness, and hospital length of stay are compared.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients between the ages of 19 and 70 undergoing total hip arthroplasty under spinal anesthesia
* Be able to provide written consent to participate in clinical trials, understand the procedures of this clinical trial, and be able to properly fill out patient-reported questionnaires
* ASA physical status classification 1-2

Exclusion Criteria:

* ASA physical status classification 3-4
* Patients who are contraindicated to nerve blocks (hypersensitivity to local anesthetics, infection at the injection site, etc.)
* Patients with chronic pain and taking pain medications, antidepressants, and anticonvulsants
* Other major medical or psychiatric conditions that will affect response to treatment
* Refusal of intravenous patient-controlled analgesia
* Patients determined to be unsuitable for this clinical trial by the researchers

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2022-10-21 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Total opioids use for 24 hours | Over the first 24 hours after surgery
  Total dose of opioids used upto 24 hours after surgery (morphine milligram equivalents)

SECONDARY OUTCOMES:
Postoperative pain at rest (Numeric rating scale) | At postoperative 4, 8, 12, 16, 20, 24 hours
  Postoperative pain at rest (Numeric rating scale; minimum 0, maximum 10, a higher score means more pain)
Postoperative pain with movement (Numeric rating scale) | At postoperative 4, 8, 12, 16, 20, 24 hours
  Postoperative pain with movement (Numeric rating scale; minimum 0, maximum 10, a higher score means more pain)
Time to first request for pain medication | From the end of surgery to discharge, an average of 4 days
  Time to first request for pain medication after surgery
Incidence of postoperative nausea and vomiting | Over the first 24 hours after surgery
  Incidence of postoperative nausea and vomiting (%)
Patient satisfaction score with pain control at 24 hours after surgery | At 24 hours after surgery
  Patient satisfaction score with pain control at 24 hours after surgery (minimum 0, maximum 10, a higher score means higher satisfaction)
Quality of Recovery at 24 hours after surgery | At 24 hours after surgery
  Quality of Recovery at 24 hours after surgery assessed by QoR-15 questionnaire
Time to discharge readiness | From the end of surgery to discharge, an average of 4 days
  Days of hospitalization after surgery until discharge readiness (defined as satisfying the following three criteria; (1) adequate pain control (numeric rating scale score < 4), (2) no intravenous opioid use in the past 12 hours, and (3) able to walk at least 30 m without time limit)
Hospital length of stay | From the end of surgery to discharge, an average of 4 days
  Days of hospitalization after surgery until discharge

CONTACTS AND LOCATIONS:
Overall Officials: Seokha Yoo, M.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No